CLINICAL TRIAL: NCT04999475
Title: Evaluation of the Effectiveness of Robotic Assisted Ultrasonography System (ROBUST) in the Clinical Environment.
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Collaborators: Sengkang General Hospital (Other); Servo Dynamics (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019/2491
Record Dates: First submitted 2021-07-22; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Abdominal Ultrasound Scanning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Work-related musculoskeletal disorders (WRMSD) among sonographers/radiographers are prevalent in the healthcare industry. This study will evaluate the use of a robotic assisted ultrasonography system (ROBUST) against the conventional abdominal ultrasound scanning procedure. The ROBUST will be developed to provide 6 degrees of freedom to allow radiographers to perform abdominal scanning without having to reach over patients. 6 sonographers with at least 5 years of experience will be recruited from SGH and SKH, to perform abdominal ultrasound scans on 50 patients. Patients will be screened by the radiographers in the study team for their suitability in the participation during their scheduled appointments and will be invited to undergo scanning with the ROBUST upon agreement. Outcome measures will include ultrasound image quality, sonographer feedback and comfort level as well as satisfaction feedback from patients. A panel of 4 reviewers, consisting of 2 radiologists and 2 senior radiographers will be invited to grade the images, using a 3-point Likert scale to compare the images taken with ROBUST against the images taken conventionally prior to using the ROBUST. The duration of each session will be recorded. The comfort level reported by sonographers will be assessed using the SGH Comfort Level Survey. In addition, the comfort level of participating patients will also be assessed using a satisfaction questionnaire. The investigators hypothesize that there is no difference in imaging quality and comfort levels of sonographers and patients between a conventional ultrasound scan and scanning with the ROBUST. The investigators also hypothesize that there would be a reduction in the risk of WRMSD among sonographers with reduction in ergonomic risk factors.

DETAILED DESCRIPTION:
6 participating sonographers will be recruited from SGH and SKH to perform abdominal ultrasound scanning. 50 patients of average body habitus with BMI <30, abdominal circumference <102cm, of whom are able to ambulate independently will be screened for suitability during their scheduled appointments and recruited. These patients from SGH and SKH, will be referred by their radiographers for the study and will be screened by the Study Team Radiographers to obtain consent. Suitable patients for the study are determined after the scheduled abdominal scans are performed at the clinic.

Patients will undergo scanning with participating sonographers using the ROBUST after completion of their scheduled conventional scans. The same ultrasound scanner and probe type will be used on all participating patients by all sonographers.

At the end of both scans, participating sonographers will be required to complete a survey on comfort level. At the end of both scans, patients will be required to complete a survey on satisfaction level. The quality of the images from both scans will be graded by 4 readers: 2 consultant radiologists and 2 senior radiographers. A photometer will be used to ensure all graders interpret the images directly from a designated monitor under consistent lighting condition.

In the first stage, ROBUST intends to scale up to expand across SingHealth institutions via a commercial partner. Together with the team, the company will engage key opinion leaders, key stakeholders and key users of respective healthcare institutions in Singapore. The team will work closely with the identified deployment partners to develop customised solutions to suit specific requirements based on disease and type of ultrasound services provided by the healthcare institutions. If successful, the ROBUST can be deployed in all ultrasound examination rooms to benefit larger population of ultrasound radiographers in managing manpower limitation and reducing work-related musculoskeletal risks. ROBUST is designed to be universal and can integrate with existing ultrasound probe, eliminating the need for a new capital purchase.

In the second stage, ROBUST will further be deployed to other national healthcare cluster within Singapore. To achieve stage 1 and stage 2 of deployment plan, the ROBUST project team will seek endorsement from key stakeholders of healthcare clusters, Group CEOs and Group COOs from NHG and NUHS at the national level to encourage technology adoption by the respective healthcare clusters.

Following success of stage 1 and stage 2, ROBUST will be marketed to key regions in Asia and Pacific countries especially ageing population nations like Japan, Hong Kong, South Korea, Australia and New Zealand through strategic distribution partners. In the third stage, based on a universal platform, ROBUST can be further expanded into the surgical domain to enable assistive solution to surgeons operating in long duration. Similarly, ROBUST can help to mitigate risk of musculoskeletal disorders among surgeons and doctors.

ELIGIBILITY:
Inclusion Criteria:

Sonographer:

-Experienced sonographers/ radiographers with more than 5 years of experience

Patient:

* BMI <30
* Abdominal circumference <102cm
* Independent Ambulation

Exclusion Criteria:

Sonographer:

-With previously reported work-related or non-work related musculoskeletal discomfort or injury

Patient:

* Pregnancy
* Non-compliance/difficulty in adhering to instructions (e.g. control breathing)
* No known muscular disorders

Ages: 21 Years to 80 Years
Age Groups: Adult, Older Adult
Study Population: Inpatients and Outpatients of Singapore General Hospital undergoing abdominal ultrasound scanning.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Comparing Quality / Grading of ultrasound image for manual scanning and robot scanning | through recruitment completion, an average of 3 months
Comparing comfort level from sonographers for manual scanning and robot scanning | through recruitment completion, an average of 1 month
Comparing satisfaction level of patients for manual scanning and robot scanning | after scanning completion, after 40 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore